CLINICAL TRIAL: NCT00311909
Title: Thalamic Deep Brain Stimulation for Tourette Syndrome: A Prospective Clinical Trial
Brief Title: Thalamic Deep Brain Stimulation for Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UHC DBS TS
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; Deep Brain Stimulation; Video assessment; YGTSS; TSSL
MeSH Terms: conditions — Tourette Syndrome

INTERVENTIONS:
Device: Thalamic deep brain stimulation

SUMMARY:
The purpose of this study is to determine whether deep brain stimulation is effective at reducing tic frequency and severity in adults with Tourette syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* Diagnosis of Tourette Syndrome by DSM-IV
* Tic frequency at least one per minute at screening
* prior failure of at least two dopamine receptor or presynaptic blockers
* negative impact on quality of life

Exclusion Criteria:

* significant structural brain lesion (on imaging studies)
* significant dementia
* severe head trauma preceding onset of tics
* use of dopamine receptor blockers prior to recognition of tics
* prior implanted electrical device
* electroconvulsive therapy (ECT) within 24 months
* suicide attempt within 12 months
* significant sociopathic personality
* current or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
modified Rush Video Rating Scale (mRVRS)

SECONDARY OUTCOMES:
tic counts (on video recording)
Yale Global Tourette Severity Scale (YGTSS)
Tourette Syndrome Symptom List (TSSL)
Quality of Life Visual Analog Scale (VAS)
SF-36
Neuropsychological battery

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Maciunas, MD MPH FACS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States